CLINICAL TRIAL: NCT03862404
Title: Double-blind Comparison of Intrapleural Bupivacaine and Saline for Ipsilateral Shoulder Pain After Thoracotomy in Patients Receiving Thoracic Epidural Analgesia
Brief Title: Intrapleural Bupivacaine for Ipsilateral Shoulder Pain After Thoracotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, JF Asenjo, Professor of Anesthesia, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-3277
Record Dates: First submitted 2019-02-19; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Post Thoracic Surgery
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: RCT with one active group and a control (placebo) group
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinded drug preparation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Patients in this group receive Normal Saline injection in the inter pleural space
  Interventions: Drug: Normal saline
- Experimental group (Experimental): Patients in this group receive Bupivacaine 0.25% + Epinephrine 5 mcg/ml injection in the inter pleural space
  Interventions: Drug: Bupivacaine-epinephrine

INTERVENTIONS:
Drug: Bupivacaine-epinephrine — See previous description
  Arms: Experimental group
Drug: Normal saline — See previous descreption
  Arms: Control group

SUMMARY:
While thoracic epidural could control incisional pain after thoracotomy, an excruciating ipsilateral shoulder pain happens post thoracotomy and could affect up to 85% of thoracotomy patients. It is often difficult to manage and relatively resistant to opioids. The investigators postulate that in the presence of a functioning thoracic epidural, intrapleural bupivacaine administered through the chest tube could be effective in reducing post thoracotomy ipsilateral shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female, between 18 and 80 years, ASA 1-3, Scheduled for open thoracotomy

Exclusion Criteria:

* ASA >3, morbid obesity BMI>40, Previous cardiac or ipsilateral thoracic surgery, Renal or hepatic failure, anemia, allergy to local anesthetics, contraindications to receive regional anesthesia, patient refusal, reiteration due to complication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Change in VAS scores | from 0 hour to 24 hour
  ISP visual analogue scale scores before intrapleural block and at 30 min, 4 hours and 24 hours

SECONDARY OUTCOMES:
Forced Vital Capacity | from 0 hour to 48 hour
Total epidural infusion | from 0 hour to 48 hour
Co-analgesia consumption | from 0 hour to 48 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided